CLINICAL TRIAL: NCT00284596
Title: Fixation Stability and Progress of Bony Healing Following Open-Wedge High- Tibial Osteotomy A 24-Subject Clinical Pilot Study Using Radio Stereometric Analysis
Brief Title: Fixation Stability and Bony Healing Following Open Wedge High Tibial Osteotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fowler Kennedy Sport Medicine Clinic (Other)
Responsible Party: Robert Giffin, FKSMC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10268
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Opening Wedge High Tibial Osteotomy
Keywords: Opening wedge high tibial osteotomy; Radio Sterometric Analysis; Locking screw fixation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: High tibial osteotomy — HTO
  Other Names: open wedge

SUMMARY:
Patients undergoing opening wedge high tibial osteotomy (HTO) will be randomized to standard or locking screw fixation of the osteotomy plate. Tantalum beads will be implanted around the osteotomy site in all subjects to facilitate RSA imaging which will then allow micromotion at the osteotomy site to be quantified.

Primary Objectives and Hypothesis

1. a)to determine fixation stability of the Puddu opening wedge osteotomy plate secured with non-locking compared to locking screws. We hypothesize that plate fixation with locking screws will result in a significant reduction of micromotion between tibial segments prior to bony healing compared to the non-locking screw fixation.

   b)To determine the progress of bony healing. We hypothesize that increased fixation stability in patients with locking screws will facilitate early bone healing reflected by smaller micromotion over time compared to the non-locking screw patients.
2. a)If there is improved stability with the use of locking screws, rehabilitation protocols following opening wedge HTO will be modified accordingly. We hypothesize that decreasing micromotion will reach the detection limit of the RSA setup (0.4 mm) earlier in the locking screw group than in the non-locking screw group.

   b)To evaluate the effect of the osteotomy on proximal tibial anatomy. We hypothesize that an open-wedge procedure might increase rather than decrease the tibial slope.

DETAILED DESCRIPTION:
For this pilot study, a total of 24 patients scheduled for opening wedge HTO who meet the inclusion criteria, have read the study letter of information and signed the informed consent will be randomized to osteotomy plate fixation with either non-locking screws (12 subjects) or locking screws (12 subjects). See flow chart 1.

Pre-operative Assessment

All subjects will undergo routine pre-operative assessment for opening wedge high tibial osteotomy which includes:

* Documentation of demographic data and medical history
* Subjective assessment of knee function using the Knee Injury and Osteoarthritis Outcome Score (KOOS)(11)
* Standard physical evaluation of the lower limb assessing range of motion, alignment, knee-related signs and symptoms
* Radiographs: standing anteroposterior hip-to-ankle;(2) lateral view; skyline patellar view at 30° of knee flexion; bilateral weight-bearing posteroanterior (PA) tunnel view at 45° of knee flexion
* Radiographic classification of arthrosis using the Kellgren scale(4)
* Measurements of mechanical and anatomical axes of the lower limb and calculation of proposed correction angles

Surgery In the operating room all subjects will undergo the following steps.

* Induction of general anaesthesia
* Percutaenous insertion into the proximal tibia surrounding the proposed osteotomy site under fluoroscopic guidance of 6 to 9 radio-opaque 0.8mm tantalum beads using a specifically designed gun. A standardized pattern of widespread tantalum bead distribution will be used. To avoid bead loosening caused by postoperative bone resorption, they will be placed a distance of at least 0.5 cm from the osteotomy line.
* RSA imaging to evaluate bead position
* Standard opening wedge HTO with the only variable being locking or non-locking screw fixation of the Puddu plate according to the randomization schedule. This procedure is routinely carried out under fluoroscopic and or radiographic control
* Second RSA imaging to obtain a reference film to assess stability
* Standard wound closure and application of hinged brace

Postoperative Treatment All subjects will undergo the routine opening wedge HTO post-operative rehabilitation protocol.

Follow-up Visits The times, number and content of follow-up visits for study subjects will not differ from the standard post-operative visits scheduled for all patients who have undergone HTO. However, because RSA imaging is specialized, this will be done at LHSC University Campus rather than at the Fowler Kennedy Sport Medicine Clinic (FKSMC). This will be communicated to patients in the letter of information. Study follow-up visits are at 2, 6,12 weeks, and 6 months after surgery.

At each study follow-up visit subjects will undergo:

* A subjective assessment of knee function using the KOOS
* A standard physical evaluation of the lower limb assessing range of motion, alignment, knee-related signs and symptoms
* Radiographs: standing anteroposterior hip-to-ankle
* RSA imaging in the AP and lateral planes simultaneously

Radiographs from each follow-up visit will be evaluated for classification of arthrosis using the Kellgren scale(4) and for measurements of mechanical and anatomical axes of the lower limb and calculation of the correction angle obtained with HTO. Translations between tibial segments will be calculated as previously described on the RSA images

ELIGIBILITY:
Inclusion Criteria:

* All patients between the ages of 30 and 70 years of age scheduled for HTO
* Localized, activity-related knee pain· Varus alignment
* Medial unicompartmental degenerative osteoarthritis
* No significant patellofemoral symptoms
* A ligamentously stable knee
* Fixed flexion of <5°

Exclusion Criteria:

* Advanced patellofemoral osteoarthritis
* Osteoarthritic involvement of the lateral compartment
* A decreased range of motion less than 90° and a flexion deformity that exceeds 10°
* Knee ligament instability
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, that would interfere with adherence to study requirements
* Serious illness (requiring systemic treatment and/or hospitalization) until subject either completes therapy or is clinically stable on therapy
* Inability of patient to speak, read or understand English
* Inability or unwillingness of subject or legal guardian/representative to give written informed consent.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-02; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The primary outcomes are the fixation stability of the implant | 2 years

SECONDARY OUTCOMES:
Validated disease specific outcome measures | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Giffin, MD, Principal Investigator — The University of Western Ontario
Locations (1):
- Fowler Kennedy Sport Medicine Clinic, University of Western Ontario, London, Ontario, Canada